CLINICAL TRIAL: NCT03897426
Title: Image Based Mobile System for Dietary Assessment and Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrent Health (Industry)
Collaborators: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HHSN261201400053C_SBIR 308
Record Dates: First submitted 2017-12-31; First posted 2019-04-01 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care arm (No Intervention): Patients randomized to the Standard-of-care-arm were provided 60 minutes of RD time for consultation through in person visits.
- Intervention arm (Experimental): Mediterranean Diet - Remote Coaching using a Mobile App.
  Patients randomized to the intervention arm were allotted 60 minutes of RD time through a Mobile App (for remote consultation), given an instruction booklet on using Mobile App, directed to a website for additional instruction on its use, and have the app set up to establish connectivity to the RD. Remote coaching by RD was the intervention.
  Interventions: Behavioral: Mediterranean Diet - Remote Coaching using a Mobile App

INTERVENTIONS:
Behavioral: Mediterranean Diet - Remote Coaching using a Mobile App — Patients randomized to the intervention arm will be then given an instruction booklet on using Mobile App, directed to a website for additional instruction on its use, and have the app set up to establish connectivity to the RD.
  Arms: Intervention arm

SUMMARY:
Vignet partnered with The George Washington University Hospital to conduct a randomized control trial (RCT) with to evaluate the system's potential to improve health outcomes for patients with CVD. Results from the RCT have the potential to be applied to patients in other chronic disease contexts.

DETAILED DESCRIPTION:
84 million American adults (>1 in 3) have cardiovascular disease, and cardiovascular disease accounts for 1 of every 3 deaths in the United States and has been the number one cause of deaths in every year since 1918. In addition, strokes, heart attacks, and uncontrolled hypertension are sources of significant disability. However, with control of known cardiovascular risk factors (i.e., smoking, body mass index, physical activity, healthy diet, total cholesterol, blood pressure, fasting plasma glucose), the risk of developing cardiovascular disease is markedly reduced. The most uncontrolled risk factor of these seven metrics for cardiovascular health amongst US adults is healthy dietary behaviors. 73 percent of Americans have a poor diet, and <1 percent have an ideal diet. No other metric of cardiovascular risk comes close - by comparison, the second worst metric is body mass index for which 31 percent have an ideal score, and the remaining five risk factors are all greater than 40 percent with ideal control. The magnitude of the gap that needs closure is greatest with healthy dietary behaviors, yet it frequently receives the least amount of intervention, and the gap has worsened over the past quarter century. Fewer patients with hypertension today are adhering to healthy nutritional habits than patients a quarter century ago. These suboptimal dietary habits are the leading cause of mortality and disability-adjusted life-years lost, greater than smoking, obesity, physical inactivity, high cholesterol, hypertension, or diabetes.

Lifestyle modification is the cornerstone of cardiovascular disease prevention, and healthy nutritional habits are essential to reducing cardiovascular risk. Changes in diet alone are as effective as blood pressure medications, without side effects associated with pharmacologic intervention. Increase nut consumption lowers cholesterol, and reducing sugar-sweetened beverages reduces risk of weight gain.

More recently, greater attention has been brought to the Mediterranean diet. The Mediterranean diet lowers blood pressure, increases HDL cholesterol, and decreases glucose levels. The term "Mediterranean diet" was first coined by Ancel Keys, best known for the Seven Countries Study, which found lower cardiovascular mortality in Mediterranean vs. non-Mediterranean countries. Since Keys' seminal work, multiple observational studies and randomized controlled trials have demonstrated a diet characterized by abundant olive oil and nut consumption and enriched for fruits, vegetables and fatty fish to be the most likely to reduce risk of cardiovascular events, including myocardial infarction, stroke and death. The Mediterranean diet was speculated to have cardiovascular benefit after observational studies suggested benefit, and the evidence solidified after randomized controlled studies showed superiority of the Mediterranean diet in both high-risk primary prevention populations and secondary prevention populations. The PREDIMED study showed a 30 percent reduction in major adverse cardiovascular events, largely through a reduction in stroke, for those patients at high risk for the development of atherosclerotic disease on a Mediterranean diet enriched for olive oil and nut consumption. The Lyon Diet Heart Study enrolled patients after a first myocardial infarction, and those randomized to receiving a Mediterranean diet enriched with more bread, fish, root vegetables and fish had improved survival and fewer myocardial infarctions than those on a usual prudent diet. Neither study demonstrated any adverse effects of the diet. These studies, however, were conducted in Mediterranean countries, and whether this diet can be successfully implemented in a non-Mediterranean population (and whether the benefits would similarly translate) remains to be tested. Observational studies suggest its possibility in a non-Mediterranean population but this finding remains to be confirmed by randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients with ongoing cardiology care with a cardiologist based at the GWU MFA and are expected to remain in the care of that cardiologist for at least 6 months.
2. Patients must own their own Android- or Apple iOS-based smartphone with a data plan.
3. Patients must give informed consent.
4. English language requirement.
5. At least 5th grade literacy level as assessed with Rapid Estimate of Adult Literacy in Medicine (REALM).[ ]
6. Patients must demonstrate an ability to download and install the Vignet FitNinja app.
7. Patient must be at least 18 years of age.
8. Patient with evidence of prior acute coronary syndrome, history of myocardial infarction, stable or unstable angina, coronary or other arterial revascularization, ischemic non-embolic stroke/TIA, or peripheral artery disease presumed to be of atherosclerotic origin.
9. Patient is on optimal medical therapy as determined by the primary cardiologist at time of enrollment.

Exclusion Criteria:

1. Clinical instability at time of enrollment.
2. Co-morbid medical disease that would preclude ability to participate in a nutrition intervention study (e.g., digestive disease with fat intolerance, life expectancy less than 5 years, severe neurologic, psychiatric or endocrine abnormalities).
3. Immunodeficiency or HIV-positive status.
4. Illegal drug use, alcoholism or daily alcohol intake >80 g/d.
5. BMI>40 kg/m2.
6. Inability or unwillingness to change dietary habits as predicted by the Prochaska and DiClemente stages of change model.[ ]
7. Inability or unwillingness to adhere to a Mediterranean diet (e.g., religious/moral reasons, disorders or chewing or swallowing).
8. Allergies to major components of the Mediterranean diet (i.e., nuts, olive oil).
9. Participation in any drug trial or use of any investigational drug within the past one year.
10. Patients who are institutionalized, lack autonomy, are non-ambulatory, lack a stable address, or have a history of missing more than one appointment in the past 6 months.
11. Patients with an acute infection or inflammation (e.g., pneumonia) in the past 3 months.
12. Pregnancy.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Compare the Mediterranean Diet Compliance Score at 3 months between the intervention and standard of care groups | 3 months
  The primary endpoint is to compare the Mediterranean Diet Compliance Score, on a scale of 0 to 14, at 3 months between the intervention and standard of care groups. Basic comparisons will be made using Wilcoxon tests to compare medians between the two groups with repeated measures analysis of variance used to compare differences across groups and over time. The higher value represents a better outcome. Subscales will not be combined.
Compare the Mediterranean Diet Compliance Score at 6 months between the intervention and standard of care groups | 6 months
  The primary endpoint is to compare the Mediterranean Diet Compliance Score, on a scale of 0 to 14, at 6 months between the intervention and standard of care groups. Basic comparisons will be made using Wilcoxon tests to compare medians between the two groups with repeated measures analysis of variance used to compare differences across groups and over time. The higher value represents a better outcome. Subscales will not be combined.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi BG, Dhawan T, Metzger K, Marshall L, Akbar A, Jain T, Young HA, Katz RJ. Image-Based Mobile System for Dietary Management in an American Cardiology Population: Pilot Randomized Controlled Trial to Assess the Efficacy of Dietary Coaching Delivered via a Smartphone App Versus Traditional Counseling. JMIR Mhealth Uhealth. 2019 Apr 23;7(4):e10755. doi: 10.2196/10755. PMID 31012860